CLINICAL TRIAL: NCT02483741
Title: The Effect of Topical Application of Manuka Honey on Healing After Extraction of Impacted Lower Third Molars: A Split-Mouth Design Randomized Controlled Trial
Brief Title: The Use of Manuka Honey to Improve Healing After Third Molars Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-OMFS-04-2015
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Surgical Extraction of Impacted Third Molars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manuka Honey (Experimental): Manuka Honey will be placed in the sockets of the extracted third molars in this group
  Interventions: Biological: Manuka Honey
- Traditional Extraction (No Intervention): No any special material will be placed in the sockets of the extracted third molars in this group

INTERVENTIONS:
Biological: Manuka Honey — This material is going to be placed into the sockets of the extracted third molars in the experimental group
  Arms: Manuka Honey

SUMMARY:
Since there is an evidence that Manuka honey is an antibacterial agent, the present study aims to confirm this characteristic and assess its effect in improving healing and reducing postsurgical symptoms, if topically applied after the surgical removal of impacted mandibular third molars

DETAILED DESCRIPTION:
Sufficient evidence exists recommending the use of honey in the management of acute wounds and burns. Studies revealed that the healing effect of honey could be classified by its antibacterial, antiviral, anti-inflammatory and antioxidant properties of its components. Manuka honey has been shown to inhibit a wide range of microorganisms, including multiresistant strains. This unique honey is derived from flowers of manuka tree (Leptospermum scoparium) in New Zealand. Dihydroxyacetone and methylglyoxal are unique and naturally occurring constituents of manuka honey that correlate with its antibacterial activity.

Since surgical extraction of impacted molars is one of the most common operations in the oral cavity and the postoperative symptoms disturbing the patient may reduce the quality of health service, this study aims to assess the healing potential of Manuka honey in reducing these symptoms by comparing the outcome of extraction of impacted lower molars with and without topical application of Manuka honey into the extraction socket.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic, Symmetrical, Bilateral Impacted Third Molars

Exclusion Criteria:

* Uncontrolled diabetes,
* Hypersensitivity to Honey
* Alcoholism,
* Drug abuse,
* Pathological condition in the region

Ages: 20 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Levels of postoperative discomfort | 7 days after the surgical removal of third molars
  Postoperative Symptom Severity (PoSSe) Scale will be used for this variable. The patient will be asked to fill in a questionnaire on the 7th day following surgery. This questionnaire is used to assess postoperative discomfort in patients who have third molars extracted. PoSSe Scale consists of 7 sub-scales that investigate the patient's ability to enjoy food; speak properly; perceive altered sensations, appearance, pain, and sickness; and interference with daily activities.
Change of facial contours due to swelling | Measurements will be taken before surgery, on the 3rd and on the 7th days after surgery.
  In order to assess facial swelling, the distances between the labial commissure and the tragus, and between the lateral canthus and the gonion will be measured.
  The change between 3 days and before surgery will give an idea about the amount of swelling that occurred following surgery.
  Between 3 days and 7 days will give an idea about the change that occurred in this period.
Change of the masticatory muscles status | Measurements will be taken before surgery, on the 3rd and on the 7th days after surgery.
  Mouth opening range will be assessed by measuring the distance between the upper and lower incisors using a vernier caliper when the patient is asked to open his/her mouth as much as possible.
  The presence of limited opening of the mouth is an indication of trismus.
Pain and Change of pain | This will be assessed on the 3rd and 7th day following surgery
  using a Visual Analog Scale of Faces (VASoF).
The presence or absence of alveolar osteitis | This will be assessed on the 3rd and 7th day following surgery
  The presence of a dry socket condition will be checked out at two time points.

SECONDARY OUTCOMES:
Time required to hemostasis | This will be recorded by the patient in the immediate postsurgical phase (i.e. between 10 minutes up to 72 hours following surgery)
Bone density and quality | at six months following surgery
  This will be assessed using Cone-beam computed tomography (CBCT) images. Hounsfield Units will be used to quantify bone density and quality.
Change of bone healing status | at 3 and six months following surgery
  This will be assessed using panoramic radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Nuraldeen Al-Khanati, DDS, Principal Investigator — MSc student, Oral and Maxillofacial Department, University of Damascus Dental School; Yasser Al-Moudallal, DDS MSc PhD, Study Director — Associate Professor of Oral and Maxillofacial Surgery, University of Damascus Dental School
Locations (1):
- Department of Oral and Maxillofacial Surgery, University of Damascus Dental School, Damascus, Damscus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atrott J, Haberlau S, Henle T. Studies on the formation of methylglyoxal from dihydroxyacetone in Manuka (Leptospermum scoparium) honey. Carbohydr Res. 2012 Nov 1;361:7-11. doi: 10.1016/j.carres.2012.07.025. Epub 2012 Aug 8. PMID 22960208
- [Background] Mavric E, Wittmann S, Barth G, Henle T. Identification and quantification of methylglyoxal as the dominant antibacterial constituent of Manuka (Leptospermum scoparium) honeys from New Zealand. Mol Nutr Food Res. 2008 Apr;52(4):483-9. doi: 10.1002/mnfr.200700282. PMID 18210383
- [Background] Rathnam A, Madan N, Madan N. The language of pain: A short study. Contemp Clin Dent. 2010 Jul;1(3):142-5. doi: 10.4103/0976-237X.72778. PMID 22114404
- [Background] Ruta DA, Bissias E, Ogston S, Ogden GR. Assessing health outcomes after extraction of third molars: the postoperative symptom severity (PoSSe) scale. Br J Oral Maxillofac Surg. 2000 Oct;38(5):480-7. doi: 10.1054/bjom.2000.0339. PMID 11010778
- [Background] Singh V, Pal US, Singh R, Soni N. Honey a sweet approach to alveolar osteitis: A study. Natl J Maxillofac Surg. 2014 Jan;5(1):31-4. doi: 10.4103/0975-5950.140166. PMID 25298714
- [Background] Wijesinghe M, Weatherall M, Perrin K, Beasley R. Honey in the treatment of burns: a systematic review and meta-analysis of its efficacy. N Z Med J. 2009 May 22;122(1295):47-60. PMID 19648986
- [Background] Yaghoobi R, Kazerouni A, Kazerouni O. Evidence for Clinical Use of Honey in Wound Healing as an Anti-bacterial, Anti-inflammatory Anti-oxidant and Anti-viral Agent: A Review. Jundishapur J Nat Pharm Prod. 2013 Aug;8(3):100-4. doi: 10.17795/jjnpp-9487. Epub 2013 Jul 17. PMID 24624197